CLINICAL TRIAL: NCT04129723
Title: Stopping Biological Therapy in Perianal Crohn's Disease Patients With Radiologically Healed Fistulas: a Prospective Cohort Study
Brief Title: Stopping Biological Therapy in PCD Study
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: No suitable case identified
Sponsor: Chinese University of Hong Kong (Other)
Responsible Party: Principal Investigator, Mak Wing Yan, Assistant Professor, Chinese University of Hong Kong
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: STOP-PCD
Record Dates: First submitted 2019-10-15; First posted 2019-10-17 (Actual); Last update posted 2022-01-28 (Actual); Status verified 2022-01

CONDITIONS: Perianal Crohn Disease; MRI; Biological Therapy
Keywords: pCD

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Perianal Crohn's patient (Experimental): Stopping biological therapy
  Interventions: Other: Stopping biological therapy

INTERVENTIONS:
Other: Stopping biological therapy — Stopping biological therapy The primary endpoint is clinical relapse at 12 months

SUMMARY:
The purpose of this which studied the biological therapy can be safely withdrawn in perianal Crohn's disease patients with radiologically healed fistula on MRI pelvis.

DETAILED DESCRIPTION:
This clinical trial in perianal Crohn's disease patients with radiologically healed fistula on MRI pelvis which studied the biological therapy can be safely withdrawn.

The primary endpoint is clinical relapse at 12 months.

ELIGIBILITY:
Inclusion Criteria:

* 1. At least 18 years old 2. Have a confirmed diagnosis of perianal Crohn's disease according to established clinical, endoscopic, radiological and histologic criteria 3. On biological therapy (anti-tumour necrosis factor, anti-integrin, anti-IL12/23) for at least 6 months 4. Confirmation of radiologically healed perianal Crohn's fistulas on MRI pelvis within the past 12 months by experienced radiologists 5. In steroid-free clinical remission for at least 6 months with fecal calprotectin <250 μg/g 6. Stable doses of immunosuppressants for at least 3 months if immunosuppressants are used 7. Written informed consent

Exclusion Criteria:

* 1. History of severe acute or delayed infusion reaction to biological therapy 2. Fistulising Crohn's disease to organs other than perianal Crohn's fistula (fistulation to skin, intestines, bladder etc.) 3. Prior history of diverting ileostomy, colostomy, proctocolectomy or proctectomy 4. Known pregnancy 5. Terminal illness

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2022-01-01 (Estimated); Primary Completion 2023-12-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Rate of perianal Crohn's disease relapse within 12 months after stopping | 12 months
  Relapse rate of patient will be calculated

SECONDARY OUTCOMES:
Rate of luminal Crohn's disease relapse within 12 months after stopping biological therapy | 12 months
  Relapse rate of patient will be calculated
Efficacy of re-treatment with biological therapy after luminal Crohn's disease relapse | 12 months
  Relapse rate of patient will be calculated
Factors associated with relapse of perianal Crohn's disease after stopping biological therapy | 12 months
  Factors associated factors will be measured by questionnaire and clinical assessment
Factors associated with relapse of luminal Crohn's disease after stopping biological therapy | 12 months
  Factors associated factors will be measured by questionnaire and clinical assessment

CONTACTS AND LOCATIONS:
Overall Officials: Wing Yan Mak, MRCP, Principal Investigator — Chinese University of Hong Kong
Locations (1):
- The Chinese University of Hong Kong, Hong Kong, Hong Kong

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Mak WY, Mak OS, Lee CK, Tang W, Leung WK, Wong MTL, Sze ASF, Li M, Leung CM, Lo FH, Lam BCY, Chan KH, Shan EHS, Tsang SWC, Hui AJ, Chow WH, Chan FKL, Sung JJY, Ng SC. Significant Medical and Surgical Morbidity in Perianal Crohn's Disease: Results from a Territory-Wide Study. J Crohns Colitis. 2018 Nov 28;12(12):1392-1398. doi: 10.1093/ecco-jcc/jjy120. PMID 30165543
- [Background] Beaugerie L, Seksik P, Nion-Larmurier I, Gendre JP, Cosnes J. Predictors of Crohn's disease. Gastroenterology. 2006 Mar;130(3):650-6. doi: 10.1053/j.gastro.2005.12.019. PMID 16530505
- [Background] Sands BE, Anderson FH, Bernstein CN, Chey WY, Feagan BG, Fedorak RN, Kamm MA, Korzenik JR, Lashner BA, Onken JE, Rachmilewitz D, Rutgeerts P, Wild G, Wolf DC, Marsters PA, Travers SB, Blank MA, van Deventer SJ. Infliximab maintenance therapy for fistulizing Crohn's disease. N Engl J Med. 2004 Feb 26;350(9):876-85. doi: 10.1056/NEJMoa030815. PMID 14985485
- [Background] Colombel JF, Sandborn WJ, Rutgeerts P, Enns R, Hanauer SB, Panaccione R, Schreiber S, Byczkowski D, Li J, Kent JD, Pollack PF. Adalimumab for maintenance of clinical response and remission in patients with Crohn's disease: the CHARM trial. Gastroenterology. 2007 Jan;132(1):52-65. doi: 10.1053/j.gastro.2006.11.041. Epub 2006 Nov 29. PMID 17241859
- [Background] Yassin NA, Askari A, Warusavitarne J, Faiz OD, Athanasiou T, Phillips RK, Hart AL. Systematic review: the combined surgical and medical treatment of fistulising perianal Crohn's disease. Aliment Pharmacol Ther. 2014 Oct;40(7):741-9. doi: 10.1111/apt.12906. Epub 2014 Aug 13. PMID 25115149
- [Background] Tozer PJ, Burling D, Gupta A, Phillips RK, Hart AL. Review article: medical, surgical and radiological management of perianal Crohn's fistulas. Aliment Pharmacol Ther. 2011 Jan;33(1):5-22. doi: 10.1111/j.1365-2036.2010.04486.x. Epub 2010 Oct 29. PMID 21083581
- [Background] Ng SC, Plamondon S, Gupta A, Burling D, Swatton A, Vaizey CJ, Kamm MA. Prospective evaluation of anti-tumor necrosis factor therapy guided by magnetic resonance imaging for Crohn's perineal fistulas. Am J Gastroenterol. 2009 Dec;104(12):2973-86. doi: 10.1038/ajg.2009.509. Epub 2009 Sep 15. PMID 19755971
- [Background] Tozer P, Ng SC, Siddiqui MR, Plamondon S, Burling D, Gupta A, Swatton A, Tripoli S, Vaizey CJ, Kamm MA, Phillips R, Hart A. Long-term MRI-guided combined anti-TNF-alpha and thiopurine therapy for Crohn's perianal fistulas. Inflamm Bowel Dis. 2012 Oct;18(10):1825-34. doi: 10.1002/ibd.21940. Epub 2012 Jan 4. PMID 22223472
- [Background] Louis E, Mary JY, Vernier-Massouille G, Grimaud JC, Bouhnik Y, Laharie D, Dupas JL, Pillant H, Picon L, Veyrac M, Flamant M, Savoye G, Jian R, Devos M, Porcher R, Paintaud G, Piver E, Colombel JF, Lemann M; Groupe D'etudes Therapeutiques Des Affections Inflammatoires Digestives. Maintenance of remission among patients with Crohn's disease on antimetabolite therapy after infliximab therapy is stopped. Gastroenterology. 2012 Jan;142(1):63-70.e5; quiz e31. doi: 10.1053/j.gastro.2011.09.034. Epub 2011 Sep 22. PMID 21945953
- [Background] Reenaers C, Mary JY, Nachury M, Bouhnik Y, Laharie D, Allez M, Fumery M, Amiot A, Savoye G, Altwegg R, Devos M, Malamut G, Bourreille A, Flourie B, Marteau P, Vuitton L, Coffin B, Viennot S, Lambert J, Colombel JF, Louis E; Groupe d'Etude Therapeutique des Affections Inflammatoires du tube Digestif. Outcomes 7 Years After Infliximab Withdrawal for Patients With Crohn's Disease in Sustained Remission. Clin Gastroenterol Hepatol. 2018 Feb;16(2):234-243.e2. doi: 10.1016/j.cgh.2017.09.061. Epub 2017 Oct 7. PMID 28993262
- [Background] Domenech E, Hinojosa J, Nos P, Garcia-Planella E, Cabre E, Bernal I, Gassull MA. Clinical evolution of luminal and perianal Crohn's disease after inducing remission with infliximab: how long should patients be treated? Aliment Pharmacol Ther. 2005 Dec;22(11-12):1107-13. doi: 10.1111/j.1365-2036.2005.02670.x. PMID 16305724
- [Background] Bouguen G, Siproudhis L, Gizard E, Wallenhorst T, Billioud V, Bretagne JF, Bigard MA, Peyrin-Biroulet L. Long-term outcome of perianal fistulizing Crohn's disease treated with infliximab. Clin Gastroenterol Hepatol. 2013 Aug;11(8):975-81.e1-4. doi: 10.1016/j.cgh.2012.12.042. Epub 2013 Jan 30. PMID 23376316
- [Background] Legue C, Brochard C, Bessi G, Wallenhorst T, Dewitte M, Siproudhis L, Bouguen G. Outcomes of Perianal Fistulising Crohn's Disease Following Anti-TNFalpha Treatment Discontinuation. Inflamm Bowel Dis. 2018 May 18;24(6):1107-1113. doi: 10.1093/ibd/izy008. PMID 29733370
- [Background] Mak WY, Lung PFC, Hart A. In Patients With Perianal Crohn's Fistulas, What Are the Outcomes When 'Radiological Healing' Is Achieved? Does Radiological Healing of Perianal Crohn's Fistulas Herald the Time Point for Stopping a Biologic? J Crohns Colitis. 2017 Dec 4;11(12):1506. doi: 10.1093/ecco-jcc/jjx094. No abstract available. PMID 28981618
- [Background] Wei SC. Differences in the public medical insurance systems for inflammatory bowel disease treatment in Asian countries. Intest Res. 2016 Jul;14(3):218-23. doi: 10.5217/ir.2016.14.3.218. Epub 2016 Jun 27. PMID 27433143